CLINICAL TRIAL: NCT01472042
Title: A Prospective Evaluation Of Biomarkers Associated With Sports Induced Concussions In College Student Athletes
Brief Title: A Evaluation Of Biomarkers Associated With Sports Induced Concussions In College Student Athletes
Acronym: GATOR
Status: Completed | Type: Observational
Sponsor: Banyan Biomarkers, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ATO-07
Record Dates: First submitted 2011-09-07; First posted 2011-11-16 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Traumatic Brain Injury; Sports Concussion; Sports Injury
Keywords: Traumatic Brain Injury; Sport Concussion; Head Injury; Sports Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Athletic Injuries; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Whole Blood and Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Sports induced concussion: Exposure to sports induced concussion
  Interventions: Other: Banyan Biomarkers
- Routine Athletic Exertion: Exposure to routine athletic exertion (non-concussion control)
  Interventions: Other: Banyan Biomarkers
- Other Non-Penetrating Trauma to the Head: Exposure to other non-penetrating trauma to the head that is witnessed or self-reported
  Interventions: Other: Banyan Biomarkers

INTERVENTIONS:
Other: Banyan Biomarkers — Biomarkers to detect specific proteins.

SUMMARY:
The purpose of this study is to study the biomarkers in subjects before and after sports-induced traumatic brain injury. The assay will be studied in a sample population of subjects over the age of 18 participating in college sports.

DETAILED DESCRIPTION:
Concussion or mild traumatic brain injury (mTBI) is a condition that affects hundreds of thousands of patients worldwide. It is a biomechanically induced neurological injury, resulting in an alteration of mental status, such as confusion or amnesia, which may or may not involve a loss of consciousness. Concussion affects about 1.6 million to 3.8 million athletes yearly, most commonly in contact sports such as American football and boxing. Early clinical effects of concussion include but are not limited to behavioral changes, impairments of memory and attention, headache, unsteadiness, and rarely, catastrophic severe brain injury (sometimes described as second impact syndrome). More recently, the consequences of repetitive mTBI from multiple concussions in a sports setting are becoming evident. Repeated concussions have been associated with greater severity of symptoms, with longer recovery time, and chronically with earlier onset of age-related memory disturbances and dementia. As a result and in contradistinction to the decades-earlier perception that these injuries were benign, sports medicine professionals are now increasingly being instructed to recognize and manage concussions as soon as they occur. "Understanding the neurobiology of concussion will lead to development and validation of physiological biomarkers of this common injury." These biomarkers (e.g., laboratory tests, imaging, electrophysiology) will then allow for improved detection, better functional assessment and evidence-based return to play recommendations.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a University of Florida student athlete on a team participating in the study
* The Subject is at least 18 years of age at screening (has had their 18th birthday)
* The Subject is willing to undergo the Informed Consent process prior to enrollment into this study.
* It is the Principal Investigator's opinion that based on the knowledge of the Subject that the Subject is an appropriate candidate for the study.

Exclusion Criteria:

* Participating in another clinical study that may affect the results of either study.
* Venipuncture not feasible (i.e. skin integrity compromised at the venipuncture sites, blood vessel calcification.
* Not available for the end of season follow-up visit.
* The Subject is otherwise determined by the Investigator to be medically unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll athletes at the University of Florida, Gainesville. Teams considered for inclusion in the study are men's football, women's lacrosse and women's soccer.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2011-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in levels of TBI biomarkers from baseline | 36 months

SECONDARY OUTCOMES:
Association of TBI biomarker levels and the Post-Concussion Scale | 36 months
Association of TBI biomarker levels and the Standardized Assessment of Concussion | Baseline (beginning of Sports season), Active Phase (during Sports Season) and End of Sports Season
Association of TBI biomarker levels and the Balance Error Scoring System | 36 months
Safety | Throughout Participation in Study
  The safety endpoints include the cumulative procedure-related adverse event-free survival, and cumulative unanticipated procedure-related adverse events. The only potential risks to patients in this study are those that are normally related to routine blood collection.
Assessment of pituitary status and determination of the presence of autoantibodies. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jay Clugston, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States